CLINICAL TRIAL: NCT03736629
Title: The AZITRAMBA Trial: Azithromycin Treatment for the Airway Microbiome in Asthma
Brief Title: Azithromycin Treatment for the Airway Microbiome in Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to accrue patients, particularly after COVID pandemic.
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB17-1287
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Asthma Chronic
Keywords: Asthma; Azithromycin; Microbiome; Sputum
MeSH Terms: conditions — Asthma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): 8 weeks of placebo capsule once daily by mouth
  Interventions: Drug: Placebo
- Azithromycin (Active Comparator): 8 weeks of Azithromycin (250 mg) capsule once daily by mouth
  Interventions: Drug: Azithromycin
- Non-asthmatic controls (No Intervention): Non-asthmatic controls to assess variability of microbiome composition and diversity over time in a normal population. No intervention given.

INTERVENTIONS:
Drug: Azithromycin — 8 weeks of Azithromycin (250 mg) once daily by mouth
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study to determine whether the bacteria inside the lungs of people with asthma can be modified (changed) if they are given an antibiotic and if this change is associated with an improvement in asthma symptoms.

ELIGIBILITY:
Inclusion criteria (All participants):

1. Age 18 - 55 years
2. Able to provide informed consent
3. Smoking history < 10 pack-years

Inclusion Criteria for subjects with poorly controlled asthma

1. Methacholine PC20 < 16 mg/ml or PD 20 < 400 mcg/ml or albuterol response > 12% on FEV1 after 4 puffs of albuterol
2. Currently prescribed ICS + LABA
3. Meet definition for Th2-low asthma: peripheral blood eosinophil count < 300 and exhaled nitric oxide level < 30 ppb.

Exclusion Criteria (All participants)

1. History of allergy or intolerance to any medications used in this study
2. Medication exclusions:

   1. Current use of medications that prolong QTc interval
   2. Current use of omalizumab or other ant-IgE therapies
   3. Current use of anti-IL 5 therapies
   4. Current use of anticoagulants
3. Prednsione or other oral steroids within past 3 months
4. Pregnancy or lactation, or plans to become pregnant
5. Other respiratory or inflammatory disorders (e.g., sarcoidosis, emphysema)
6. Pre-existing liver disease by history
7. Smoking within the last 6 months
8. Exacerbation of asthma in past 3 months
9. Affected by a hearing disorder
10. Clinically significant medical condition (e.g., heart failure, seizure disorder) which may in-crease risk as determined by study investigator
11. Corrected QT interval > 450 msec. Patients with known cardiac history or prolonged QT interval on a screening EKG are excluded given the small but real potential for macrolide-related side effects

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve White, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data that is de-identified available to all qualified investigators
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon publication of the major manuscript to be generated from this study. Data will be deposited in an appropriate major database (e.g., sequencing information will be deposited in a genetics bio-bank).
Access Criteria: All qualified investigators who sign appropriate data use agreements and material transfer agreements with the University of Chicago and Northwestern University

REFERENCES:
- [Result] Vogelmeier CF, Fuhlbrigge A, Jauhiainen A, Scheepers LEJM, Bengtsson T, Peterson S, Karlsson N, Sethi T, Locantore N, Tal-Singer R, Rennard S, Fageras M, Da Silva CA. COPDCompEx: A novel composite endpoint for COPD exacerbations to enable faster clinical development. Respir Med. 2020 Nov;173:106175. doi: 10.1016/j.rmed.2020.106175. Epub 2020 Sep 28. PMID 33032168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Started | 3 | 2 | 12
Completed | 3 | 2 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls | Total
Number analyzed (Participants) | 3 | 2 | 12 | 17
Age, Continuous [Mean (Full Range); unit: years] | 50.5 [42 to 59] | 47.4 [45 to 49] | 35.5 [19 to 54] | 39.5 [19 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 9 | 14
  Male | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 5 | 8
  White | 0 | 0 | 4 | 4
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Test (ACT) Score Change From Baseline Over 8 Weeks
Description: Score ranging from 0 to 40 indicating the degree of asthma symptoms. Lower score indicating worse asthma symptoms.
Time Frame: Baseline and 8 weeks
Population: Outcome variable is not applicable to non-asthmatic controls, as they were not assessed for asthma symptoms.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 3 | 2 | 0
score on a scale | 0.67 (0.67) | 0.00 (2.00) |
Statistical Analysis 1: Comparison: Placebo vs Azithromycin; Study did not reach its accrual goal. Sample size is too small to draw any conclusions; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Net) = -0.67, 95% CI 2-sided [-6.14 to 4.81], Standard Error of Mean 1.72

2. Secondary Outcome: Forced Expiratory Volume (FEV1) Change From Baseline Over 8 Weeks
Description: Volume of air exhaled in 1 second on a forced expiration, expressed as percent of predicted, indicating the degree of airflow obstruction in asthma
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: percentage of predicted
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 3 | 2 | 12
percentage of predicted | 1.67 (3.76) | -4.00 (11.00) | -2.92 (1.37)
Statistical Analysis 1: Comparison: Placebo vs Azithromycin; Test type: Superiority; p = 0.59, t-test, 2 sided; Mean Difference (Net) = -5.67, 95% CI 2-sided [-35.98 to 24.65] — Study did not reach its accrual goal. Sample size is too small to draw any conclusions

3. Secondary Outcome: Sputum Eosinophils Change From Baseline Over 8 Weeks
Description: Percentage of 'eosinophils', an inflammatory cell seen in the airways of people with asthma, indicating the degree of inflammation
Time Frame: Baseline and 8 weeks
Population: Some patients had missing data.
Measure: Mean (Full Range); unit: percentage of eosinophils
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 1 | 1 | 5
percentage of eosinophils | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.06 [-0.33 to 0.64]

4. Secondary Outcome: Sputum Neutrophils Change From Baseline Over 8 Weeks
Description: Percentage of 'neutrophils', an inflammatory cell seen in the airways of people with asthma, indicating the degree of inflammation
Time Frame: Baseline and 8 weeks
Population: Some patients had missing data.
Measure: Mean (Full Range); unit: percentage of neutrophils
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 1 | 1 | 5
percentage of neutrophils | -0.00 [-0.00 to -0.00] | 1.59 [1.59 to 1.59] | -10.03 [-46.88 to 8.03]

5. Secondary Outcome: Number of Participants With Diary Event or Serious Asthma Exacerbation Over 8 Weeks
Description: The outcome is derived from a weighted scoring system called CompEx that describes asthma symptoms recorded on a daily basis. Final result is a dichotomous outcome indicating whether the patient had a "diary event" based on changes in peak expiratory flow, reliever use, and asthma symptoms or a serious exacerbation (deterioration of asthma leading to oral corticosteroid use, emergency room admission, or hospital admission).
Time Frame: 8 weeks
Population: Outcome measure is not applicable to non-asthmatic controls, as they were not assessed for asthma severity.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 2 | 2 | 0
Participants | 1 | 0 |
Statistical Analysis 1: Comparison: Placebo vs Azithromycin; Study did not reach its accrual goal. Sample size is too small to draw any conclusions; Test type: Superiority; p = 1.0, Fisher Exact

6. Secondary Outcome: Microbiome Shannon Alpha-diversity Score Change From Baseline to 8 Weeks
Description: A measure of the diversity of the bacteria in the sputum or oral sample; that is, how many different types of bacteria are present. This value decreases in severe asthma
Time Frame: 8 weeks
Population: Insufficient sample size for meaningful results in intervention arms due to low accrual. Microbiome assays were not performed.
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Microbiome Beta-diversity Score Change From Baseline to 8 Weeks
Description: A second measure of the diversity of the bacteria in the sputum or oral sample; that is, how many different types of bacteria are present. This value decreases in severe asthma
Time Frame: 8 weeks
Population: Insufficient sample size for meaningful results in intervention arms. Microbiome assays were not performed.
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Microbiome Change in Relative Proportion of Top 10 Genera From Baseline to 8 Weeks
Description: A measure of how many of the top types of bacteria are present in the sputum or oral sample. Value changes with asthma
Time Frame: 8 weeks
Population: Insufficient sample size for meaningful results in intervention arms. Microbiome assays were not performed.
Arm/Group | Placebo | Azithromycin | Non-asthmatic Controls
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks Note: Adverse events were not collected in the Non-asthmatic controls.
Arm/Group | Placebo | Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Azithromycin (N=2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT03736629/Prot_SAP_000.pdf